CLINICAL TRIAL: NCT06704308
Title: Development and Preliminary Evaluation of a Multilevel Intervention to Increase HPV Vaccine Confidence Among Parents of Youth in Rural KY
Brief Title: Parents' HPV Stories
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anne E Ray (Other)
Collaborators: Real Prevention, LLC (Industry); Merck Institute for Therapeutic Research (Unknown)
Responsible Party: Sponsor-Investigator, Anne E Ray, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 95632
Record Dates: First submitted 2024-11-19; First posted 2024-11-26 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: HPV Vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parents' Stories Web Application + Provider Elaborated Prompts (Experimental): Participating parents will be asked to navigate a web application that consists of (a) brief, 90-second narrative videos that encourage parent-provider communication about the vaccine and (b) personalized feedback to parents that is tailored to provide educational content in response to their concerns and be motivational in nature. Providers will provide elaborated prompts related to the vaccine when meeting with parents tailored to their concerns.
  Interventions: Behavioral: Web Application; Behavioral: Provider Elaborated Prompts

INTERVENTIONS:
Behavioral: Web Application — A web application for vaccine-hesitant parents and their teens with brief, 90-second narrative videos and tailored, motivational content
Behavioral: Provider Elaborated Prompts — A component for providers that suggests elaborated prompts to be used with parents that align with the content of the web application, are tailored to parent concerns, and are motivational in nature

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility of intervention implementation in two clinics in rural KY, and its preliminary efficacy with regards to increasing vaccine confidence in a sample of vaccine hesitant parents.

Hypothesis: Parents will report increased vaccine confidence scores post-intervention.

Data from this study will provide preliminary data for a larger scale evaluation of the intervention.

Participants will be asked to complete surveys, view a web-based intervention and then visit with their child's healthcare provider.

DETAILED DESCRIPTION:
Participants will be asked to complete a brief screening assessment to establish their eligibility for participation. Eligible participants will be asked to complete a consent form and be directed to the pre-test survey. Upon completion of the survey, the participants will be directed to the tailored intervention content, including the Parents' Stories videos. This step will be completed prior to interaction with the provider. During the provider-patient visit, the provider will deliver the elaborated prompt portion of the intervention to participating mothers. Mothers will receive a link to the post-test survey two weeks following their appointment.

ELIGIBILITY:
Inclusion Criteria:

* status as a mother or female guardian of an 11-17-year-old adolescent
* status as a U.S. resident
* self-reported ability to read English
* self-reported HPV vaccine hesitant using established methodology

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in HPV Vaccine Hesitancy Scale score | From pretest to posttest (up to two weeks)
  9-item scale from Strongly Disagree (1) to Strongly Agree (5); scores range from 1-5, with higher scores indicating greater hesitancy
Change Human Papillomavirus Knowledge Questionnaire score | From pretest to posttest (up to two weeks)
  13-item scale with True / False / I don't know response options; scores range from 0-13 with higher scores indicating greater vaccine knowledge
Change in intent to discuss HPV vaccine with provider | From pretest to posttest (up to two weeks)
  Answers include Very likely; Somewhat likely; Not too likely; Not likely at all; Not sure / do not know
Change in HPV vaccine intent | From pretest to posttest (up to two weeks)
  1 item adapted from NIS-TEEN survey. Answers include very likely; somewhat likely; not too likely; not likely at all; not sure / do not know
Change in self-reported HPV vaccination and related provider recommendations | from screening to posttest (up to two weeks)
  4 items adapted from the NIS-TEEN survey.
Change in Reasons Not to Vaccinate score | Pretest only
  16 items adapted from NIS-TEEN survey; higher score indicates more obstacles to vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Ray, PhD., Principal Investigator — University of Kentucky; Aaron Kruse-Diehr, PhD, Study Chair — University of Kentucky; Michael Hecht, PhD, Study Chair — Real Prevention, LLC
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be available to qualified researchers after the main findings are published in a peer-reviewed journal upon request. All data sharing will comply with local, state, and federal laws and regulations, including HIPAA Privacy and Security Rules. Data will be de-identified before presentations and publications, as well as any datasets shared with qualified researchers.